CLINICAL TRIAL: NCT01858649
Title: Randomized Phase 2 Study Comparing Pathological Responses on Colorectal Cancer Metastases After Preoperative Treatment Combining Bevacizumab With FOLFOX or FOLFIRI
Brief Title: Study Comparing Pathological Responses Observed on Colorectal Cancer Metastases Resected After Preoperative Bevacizumab With FOLFOX or FOLFIRI.
Acronym: BEV-ONCO2012
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Grand Hôpital de Charleroi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BEV-ONCO2012; 2012-005376-34 (EudraCT Number)
Record Dates: First submitted 2013-05-07; First posted 2013-05-21 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic; colorectal; cancer; liver; Bevacizumab; Pathological response
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — Bevacizumab; Fluorouracil; Oxaliplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Folfox: oxaliplatin +leucovorin+ 5FU (Active Comparator): FOLFOX (oxaliplatin +leucovorin+ 5FU) +bevacizumab+ metastases resection
  Interventions: Procedure: Metastases resection; Drug: Bevacizumab; Drug: 5 FU; Drug: Oxaliplatin
- FOLFIRI: irinotecan+leucovorin+5FU (Active Comparator): FOLFIRI (irinotecan+leucovorin+5FU) +bevacizumab +metastases resection
  Interventions: Procedure: Metastases resection; Drug: Bevacizumab; Drug: 5 FU; Drug: Irinotecan

INTERVENTIONS:
Procedure: Metastases resection — Surgery of colorectal cancer metastases will be proceeded after 3 to 6 cycles of chemotherapy ( folfox or folfiri) + bevacizumab .
Drug: Bevacizumab — Bevacizumab 5 mg/kg in 100 ml NaCl 0.9% IV infusion 3 to 5 cycles. No bevacizumab for ultimate cycle .
  Other Names: Avastin
Drug: 5 FU — Leucovorin L (levoleucovorin) 200 mg/m2 (or folinic acid 400 mg/m²) in 250 ml glucose 5%, IV infusion 3 to 6 cycles 5-FU bolus 400 mg/m2, IV bolus 3 to 6 cycles 5-FU continuous infusion 2400 mg/m2, 46-hour cont. IV infusion 3 to 6 cycles
  Other Names: 5-Fluorouracile
Drug: Oxaliplatin — oxaliplatin 85 mg/m² in 150 ml NaCl 0.9%, IV infusion 3 to 6 cycles
  Other Names: Eloxatin
  Arms: Folfox: oxaliplatin +leucovorin+ 5FU
Drug: Irinotecan — Irinotecan 180 mg/m² in 150 ml NaCl 0.9%, IV infusion 3 to 6 cycles
  Other Names: Campto; Irinosin
  Arms: FOLFIRI: irinotecan+leucovorin+5FU

SUMMARY:
The study is designed to analyze the pathological tumor response on resected colorectal cancer metastases after preoperative treatment with bevacizumab combined with FOLFOX or FOLFIRI regimen in a prospective cohort and to correlate this response with patient's outcome.

DETAILED DESCRIPTION:
This is a phase II , openlabel, randomized study in patients with confirmed diagnosis of resectable metastatic colorectal adenocarcinoma , who have not received prior chemotherapy for their metastatic disease. The study is designed to compare pathological responses observed after pre-operative chemotherapy bevacizumab with FOLFOX or FOLFIRI.

ELIGIBILITY:
Inclusion Criteria:

* 1. Female or male patients with at least 18 years at the time the informed consent is signed
* 2.ECOG (Eastern Cooperative Oncology Group)performance status 0 or 1
* 3.Histological or cytological confirmed diagnostic of adenocarcinoma of the colon or rectum, with or without primary tumour in situ. Wild-type or mutated KRAS tumor status.
* 4.Patients must present a resectable metastatic disease for which the decision of preoperative chemotherapy is considered. Resectability could be planned in one or multiple stage if indicated. As commonly admitted, resectability means the surgical clearance (+/- radiofrequency ablation) of all detectable (liver) lesions with tumor-free margins and compatible with an adequate hepatic reserve. Practically, bilateral tumor location, number and location of lesions, and inadequate hepatic reserve remain the main decisional factors.
* 5.Partial and minor resection of metastatic disease is allowed within 3 months before inclusion if patient has never received chemotherapy for mCRC.
* 6.Extra hepatic metastatic location is limited to 1 site. Extra-hepatic location must be easily resectable in one stage surgery.
* 7.Patients may have received adjuvant chemotherapy or (neo-) adjuvant chemo-radiotherapy to the pelvis, provided the last dose of chemotherapy was administered at least 6 months prior to inclusion (12 months for oxaliplatin). Previous radiotherapy to the pelvis is not an exclusion criterion.
* 8.Adequate haematological, renal and hepatic function as follows: Haematological Neutrophils > 1.5 x 109/L Platelets > 100 x 109/L Renal Creatinine < 1.5 x ULN (Upper Limit of Normal) Hepatic Bilirubin < 1.5 X ULN AST(Aspartate aminotransferase), ALT (Alanine Aminotransferase) < 5 x ULN Phos Alc. < 5 x ULN
* 9.Proteinuria <2+ (dipstick urinalysis) or =1g/24hour.
* 10.No history of myocardial infarction and/or stroke within 6 months prior to randomization. No uncontrolled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure > 100 mmHg), or history of hypertensive crisis, or hypertensive encephalopathy.
* 11.Female patients must either be postmenopausal, sterile (surgically or radiation- or chemically-induced), or if sexually active using an acceptable method of contraception.
* 12.Male patients must be surgically sterile or if sexually active and having a pre-menopausal partner must be using an acceptable method of contraception.
* 13.Life expectancy of at least 3 months without any active treatment.

Exclusion Criteria:

* 1.Non resectable mCRC (metastatic ColoRectal Cancer) (if resectability remains uncertain or unprobable after 3 months chemotherapy, patient is excluded from the trial).
* 2.Prior chemotherapy or systemic therapy for mCRC. Adjuvant chemotherapy for colorectal cancer is not an exclusion criterion provided that it was completed more than 6 months prior to inclusion. Oxaliplatin-based chemotherapy must be completed more than 1 year prior to inclusion.
* 3.Prior utilization of bevacizumab, aflibercept (or other anti-VEGF(vascular endothelial growth factor) therapy).
* 4.Previous radiotherapy delivered to the upper abdomen.
* 5.Evidence of ascites, cirrhosis, portal hypertension, main portal venous tumour involvement or thrombosis as determined by clinical or radiologic assessment.
* 6.Prior major liver resection: remnant liver < 50% of the initial liver volume.
* 7.Non-malignant disease that would render the patient unsuitable for treatment according to this protocol.
* 8.Concurrent central nervous systems metastases
* 9.Peripheric neuropathy ≥ grade 2.
* 10.Interstitial lung disease
* 11.Pregnant or breast feeding.
* 12.The patient has previous or concomitant malignancies, except: Invasive malignancies in remission for more than 5 years and non melanoma skin cancer or carcinoma in situ of the cervix.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
the major pathological response rate | After surgery (Metastases resection-average 3 months)
  This is at the surgery time. The metastases resection must be process after 6 cycles of randomized chemotherapy + target therapy. It depend but it will be normally 3 months after patient inclusion in the study

SECONDARY OUTCOMES:
Progression free survival | at 6 months and at 12 months after randomization
Overall Survival | At the end of the study
  The overall survival will be analyzed at the end of the study (3 years of recruitment and one years of follow-up)
Clinical Response Rate | At time of surgery - average 3 months
Metabolic Response Rate | At time of surgery - Average 3 months
Post operative complication | One month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Marc Van den Eynde, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain; Javier Carrasco, MD PhD, Principal Investigator — Grand Hôpital de Charleroi - Notre-Dame
Locations (11):
- Belgium (11):
  - Clinique Saint Luc, Bouge
  - CHIREC, Brussels
  - Cliniques universitaires Saint-Luc, Brussels
  - Grand Hopital de Charleroi, Charleroi
  - AZ Groeninge, Kortrijk
  - Centre Hospitalier Jolimont Lobbes, La Louvière
  - CHC Liège clinique Saint Joseph, Liège
  - CHU liège (Sart Timan), Liège
  - Clinique Maternité Saint Elisabeth, Namur
  - Clinique Saint Pierre Ottignies, Ottignies
  - CHU-UCL Dinant-Godinne, Yvoir

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Thun MJ. Cancer statistics, 2009. CA Cancer J Clin. 2009 Jul-Aug;59(4):225-49. doi: 10.3322/caac.20006. Epub 2009 May 27. PMID 19474385
- [Background] Jamison RL, Donohue JH, Nagorney DM, Rosen CB, Harmsen WS, Ilstrup DM. Hepatic resection for metastatic colorectal cancer results in cure for some patients. Arch Surg. 1997 May;132(5):505-10; discussion 511. doi: 10.1001/archsurg.1997.01430290051008. PMID 9161393
- [Background] Nordlinger B, Guiguet M, Vaillant JC, Balladur P, Boudjema K, Bachellier P, Jaeck D. Surgical resection of colorectal carcinoma metastases to the liver. A prognostic scoring system to improve case selection, based on 1568 patients. Association Francaise de Chirurgie. Cancer. 1996 Apr 1;77(7):1254-62. PMID 8608500
- [Background] Rees M, Tekkis PP, Welsh FK, O'Rourke T, John TG. Evaluation of long-term survival after hepatic resection for metastatic colorectal cancer: a multifactorial model of 929 patients. Ann Surg. 2008 Jan;247(1):125-35. doi: 10.1097/SLA.0b013e31815aa2c2. PMID 18156932
- [Background] Nordlinger B, Sorbye H, Glimelius B, Poston GJ, Schlag PM, Rougier P, Bechstein WO, Primrose JN, Walpole ET, Finch-Jones M, Jaeck D, Mirza D, Parks RW, Collette L, Praet M, Bethe U, Van Cutsem E, Scheithauer W, Gruenberger T; EORTC Gastro-Intestinal Tract Cancer Group; Cancer Research UK; Arbeitsgruppe Lebermetastasen und-tumoren in der Chirurgischen Arbeitsgemeinschaft Onkologie (ALM-CAO); Australasian Gastro-Intestinal Trials Group (AGITG); Federation Francophone de Cancerologie Digestive (FFCD). Perioperative chemotherapy with FOLFOX4 and surgery versus surgery alone for resectable liver metastases from colorectal cancer (EORTC Intergroup trial 40983): a randomised controlled trial. Lancet. 2008 Mar 22;371(9617):1007-16. doi: 10.1016/S0140-6736(08)60455-9. PMID 18358928
- [Background] Hurwitz H, Fehrenbacher L, Novotny W, Cartwright T, Hainsworth J, Heim W, Berlin J, Baron A, Griffing S, Holmgren E, Ferrara N, Fyfe G, Rogers B, Ross R, Kabbinavar F. Bevacizumab plus irinotecan, fluorouracil, and leucovorin for metastatic colorectal cancer. N Engl J Med. 2004 Jun 3;350(23):2335-42. doi: 10.1056/NEJMoa032691. PMID 15175435
- [Background] Saltz LB, Clarke S, Diaz-Rubio E, Scheithauer W, Figer A, Wong R, Koski S, Lichinitser M, Yang TS, Rivera F, Couture F, Sirzen F, Cassidy J. Bevacizumab in combination with oxaliplatin-based chemotherapy as first-line therapy in metastatic colorectal cancer: a randomized phase III study. J Clin Oncol. 2008 Apr 20;26(12):2013-9. doi: 10.1200/JCO.2007.14.9930. PMID 18421054
- [Background] Van Cutsem E, Kohne CH, Lang I, Folprecht G, Nowacki MP, Cascinu S, Shchepotin I, Maurel J, Cunningham D, Tejpar S, Schlichting M, Zubel A, Celik I, Rougier P, Ciardiello F. Cetuximab plus irinotecan, fluorouracil, and leucovorin as first-line treatment for metastatic colorectal cancer: updated analysis of overall survival according to tumor KRAS and BRAF mutation status. J Clin Oncol. 2011 May 20;29(15):2011-9. doi: 10.1200/JCO.2010.33.5091. Epub 2011 Apr 18. PMID 21502544
- [Background] Bokemeyer C, Van Cutsem E, Rougier P, Ciardiello F, Heeger S, Schlichting M, Celik I, Kohne CH. Addition of cetuximab to chemotherapy as first-line treatment for KRAS wild-type metastatic colorectal cancer: pooled analysis of the CRYSTAL and OPUS randomised clinical trials. Eur J Cancer. 2012 Jul;48(10):1466-75. doi: 10.1016/j.ejca.2012.02.057. Epub 2012 Mar 23. PMID 22446022
- [Background] Douillard JY, Siena S, Cassidy J, Tabernero J, Burkes R, Barugel M, Humblet Y, Bodoky G, Cunningham D, Jassem J, Rivera F, Kocakova I, Ruff P, Blasinska-Morawiec M, Smakal M, Canon JL, Rother M, Oliner KS, Wolf M, Gansert J. Randomized, phase III trial of panitumumab with infusional fluorouracil, leucovorin, and oxaliplatin (FOLFOX4) versus FOLFOX4 alone as first-line treatment in patients with previously untreated metastatic colorectal cancer: the PRIME study. J Clin Oncol. 2010 Nov 1;28(31):4697-705. doi: 10.1200/JCO.2009.27.4860. Epub 2010 Oct 4. PMID 20921465
- [Background] Khatri VP, Chee KG, Petrelli NJ. Modern multimodality approach to hepatic colorectal metastases: solutions and controversies. Surg Oncol. 2007 Jul;16(1):71-83. doi: 10.1016/j.suronc.2007.05.001. Epub 2007 May 29. PMID 17532622
- [Background] de Gramont A, Tournigand C, Andre T, Larsen AK, Louvet C. Adjuvant therapy for stage II and III colorectal cancer. Semin Oncol. 2007 Apr;34(2 Suppl 1):S37-40. doi: 10.1053/j.seminoncol.2007.01.004. PMID 17449351
- [Background] Andre T, Boni C, Mounedji-Boudiaf L, Navarro M, Tabernero J, Hickish T, Topham C, Zaninelli M, Clingan P, Bridgewater J, Tabah-Fisch I, de Gramont A; Multicenter International Study of Oxaliplatin/5-Fluorouracil/Leucovorin in the Adjuvant Treatment of Colon Cancer (MOSAIC) Investigators. Oxaliplatin, fluorouracil, and leucovorin as adjuvant treatment for colon cancer. N Engl J Med. 2004 Jun 3;350(23):2343-51. doi: 10.1056/NEJMoa032709. PMID 15175436
- [Background] Gruenberger B, Tamandl D, Schueller J, Scheithauer W, Zielinski C, Herbst F, Gruenberger T. Bevacizumab, capecitabine, and oxaliplatin as neoadjuvant therapy for patients with potentially curable metastatic colorectal cancer. J Clin Oncol. 2008 Apr 10;26(11):1830-5. doi: 10.1200/JCO.2007.13.7679. PMID 18398148
- [Background] Klinger M, Tamandl D, Eipeldauer S, Hacker S, Herberger B, Kaczirek K, Dorfmeister M, Gruenberger B, Gruenberger T. Bevacizumab improves pathological response of colorectal cancer liver metastases treated with XELOX/FOLFOX. Ann Surg Oncol. 2010 Aug;17(8):2059-65. doi: 10.1245/s10434-010-0972-9. Epub 2010 Feb 23. PMID 20177795
- [Background] Folprecht G, Gruenberger T, Bechstein WO, Raab HR, Lordick F, Hartmann JT, Lang H, Frilling A, Stoehlmacher J, Weitz J, Konopke R, Stroszczynski C, Liersch T, Ockert D, Herrmann T, Goekkurt E, Parisi F, Kohne CH. Tumour response and secondary resectability of colorectal liver metastases following neoadjuvant chemotherapy with cetuximab: the CELIM randomised phase 2 trial. Lancet Oncol. 2010 Jan;11(1):38-47. doi: 10.1016/S1470-2045(09)70330-4. Epub 2009 Nov 26. PMID 19942479
- [Background] Ribero D, Wang H, Donadon M, Zorzi D, Thomas MB, Eng C, Chang DZ, Curley SA, Abdalla EK, Ellis LM, Vauthey JN. Bevacizumab improves pathologic response and protects against hepatic injury in patients treated with oxaliplatin-based chemotherapy for colorectal liver metastases. Cancer. 2007 Dec 15;110(12):2761-7. doi: 10.1002/cncr.23099. PMID 17960603
- [Background] Kesmodel SB, Ellis LM, Lin E, Chang GJ, Abdalla EK, Kopetz S, Vauthey JN, Rodriguez-Bigas MA, Curley SA, Feig BW. Preoperative bevacizumab does not significantly increase postoperative complication rates in patients undergoing hepatic surgery for colorectal cancer liver metastases. J Clin Oncol. 2008 Nov 10;26(32):5254-60. doi: 10.1200/JCO.2008.17.7857. Epub 2008 Oct 14. PMID 18854565
- [Background] D'Angelica M, Kornprat P, Gonen M, Chung KY, Jarnagin WR, DeMatteo RP, Fong Y, Kemeny N, Blumgart LH, Saltz LB. Lack of evidence for increased operative morbidity after hepatectomy with perioperative use of bevacizumab: a matched case-control study. Ann Surg Oncol. 2007 Feb;14(2):759-65. doi: 10.1245/s10434-006-9074-0. Epub 2006 Nov 11. PMID 17103075
- [Background] Reddy SK, Morse MA, Hurwitz HI, Bendell JC, Gan TJ, Hill SE, Clary BM. Addition of bevacizumab to irinotecan- and oxaliplatin-based preoperative chemotherapy regimens does not increase morbidity after resection of colorectal liver metastases. J Am Coll Surg. 2008 Jan;206(1):96-106. doi: 10.1016/j.jamcollsurg.2007.06.290. Epub 2007 Sep 17. PMID 18155574
- [Background] Klinger M, Eipeldauer S, Hacker S, Herberger B, Tamandl D, Dorfmeister M, Koelblinger C, Gruenberger B, Gruenberger T. Bevacizumab protects against sinusoidal obstruction syndrome and does not increase response rate in neoadjuvant XELOX/FOLFOX therapy of colorectal cancer liver metastases. Eur J Surg Oncol. 2009 May;35(5):515-20. doi: 10.1016/j.ejso.2008.12.013. Epub 2009 Feb 5. PMID 19200687
- [Background] van der Pool AE, Marsman HA, Verheij J, Ten Kate FJ, Eggermont AM, Ijzermans JN, Verhoef C. Effect of bevacizumab added preoperatively to oxaliplatin on liver injury and complications after resection of colorectal liver metastases. J Surg Oncol. 2012 Dec;106(7):892-7. doi: 10.1002/jso.23142. Epub 2012 May 2. PMID 22552819
- [Background] Mandard AM, Dalibard F, Mandard JC, Marnay J, Henry-Amar M, Petiot JF, Roussel A, Jacob JH, Segol P, Samama G, et al. Pathologic assessment of tumor regression after preoperative chemoradiotherapy of esophageal carcinoma. Clinicopathologic correlations. Cancer. 1994 Jun 1;73(11):2680-6. doi: 10.1002/1097-0142(19940601)73:113.0.co;2-c. PMID 8194005
- [Background] Swisher SG, Hofstetter W, Wu TT, Correa AM, Ajani JA, Komaki RR, Chirieac L, Hunt KK, Liao Z, Phan A, Rice DC, Vaporciyan AA, Walsh GL, Roth JA. Proposed revision of the esophageal cancer staging system to accommodate pathologic response (pP) following preoperative chemoradiation (CRT). Ann Surg. 2005 May;241(5):810-7; discussion 817-20. doi: 10.1097/01.sla.0000161983.82345.85. PMID 15849517
- [Background] Ajani JA, Mansfield PF, Crane CH, Wu TT, Lunagomez S, Lynch PM, Janjan N, Feig B, Faust J, Yao JC, Nivers R, Morris J, Pisters PW. Paclitaxel-based chemoradiotherapy in localized gastric carcinoma: degree of pathologic response and not clinical parameters dictated patient outcome. J Clin Oncol. 2005 Feb 20;23(6):1237-44. doi: 10.1200/JCO.2005.01.305. PMID 15718321
- [Background] Rodel C, Martus P, Papadoupolos T, Fuzesi L, Klimpfinger M, Fietkau R, Liersch T, Hohenberger W, Raab R, Sauer R, Wittekind C. Prognostic significance of tumor regression after preoperative chemoradiotherapy for rectal cancer. J Clin Oncol. 2005 Dec 1;23(34):8688-96. doi: 10.1200/JCO.2005.02.1329. Epub 2005 Oct 24. PMID 16246976
- [Background] Bouzourene H, Bosman FT, Seelentag W, Matter M, Coucke P. Importance of tumor regression assessment in predicting the outcome in patients with locally advanced rectal carcinoma who are treated with preoperative radiotherapy. Cancer. 2002 Feb 15;94(4):1121-30. PMID 11920483
- [Background] Rubbia-Brandt L, Giostra E, Brezault C, Roth AD, Andres A, Audard V, Sartoretti P, Dousset B, Majno PE, Soubrane O, Chaussade S, Mentha G, Terris B. Importance of histological tumor response assessment in predicting the outcome in patients with colorectal liver metastases treated with neo-adjuvant chemotherapy followed by liver surgery. Ann Oncol. 2007 Feb;18(2):299-304. doi: 10.1093/annonc/mdl386. Epub 2006 Oct 23. PMID 17060484
- [Background] Blazer DG 3rd, Kishi Y, Maru DM, Kopetz S, Chun YS, Overman MJ, Fogelman D, Eng C, Chang DZ, Wang H, Zorzi D, Ribero D, Ellis LM, Glover KY, Wolff RA, Curley SA, Abdalla EK, Vauthey JN. Pathologic response to preoperative chemotherapy: a new outcome end point after resection of hepatic colorectal metastases. J Clin Oncol. 2008 Nov 20;26(33):5344-51. doi: 10.1200/JCO.2008.17.5299. Epub 2008 Oct 20. PMID 18936472
- [Background] Maru DM, Kopetz S, Boonsirikamchai P, Agarwal A, Chun YS, Wang H, Abdalla EK, Kaur H, Charnsangavej C, Vauthey JN, Loyer EM. Tumor thickness at the tumor-normal interface: a novel pathologic indicator of chemotherapy response in hepatic colorectal metastases. Am J Surg Pathol. 2010 Sep;34(9):1287-94. doi: 10.1097/PAS.0b013e3181eb2f7b. PMID 20697255
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Young H, Baum R, Cremerius U, Herholz K, Hoekstra O, Lammertsma AA, Pruim J, Price P. Measurement of clinical and subclinical tumour response using [18F]-fluorodeoxyglucose and positron emission tomography: review and 1999 EORTC recommendations. European Organization for Research and Treatment of Cancer (EORTC) PET Study Group. Eur J Cancer. 1999 Dec;35(13):1773-82. doi: 10.1016/s0959-8049(99)00229-4. PMID 10673991
- [Background] Rubbia-Brandt L, Audard V, Sartoretti P, Roth AD, Brezault C, Le Charpentier M, Dousset B, Morel P, Soubrane O, Chaussade S, Mentha G, Terris B. Severe hepatic sinusoidal obstruction associated with oxaliplatin-based chemotherapy in patients with metastatic colorectal cancer. Ann Oncol. 2004 Mar;15(3):460-6. doi: 10.1093/annonc/mdh095. PMID 14998849
- [Background] Galon J, Costes A, Sanchez-Cabo F, Kirilovsky A, Mlecnik B, Lagorce-Pages C, Tosolini M, Camus M, Berger A, Wind P, Zinzindohoue F, Bruneval P, Cugnenc PH, Trajanoski Z, Fridman WH, Pages F. Type, density, and location of immune cells within human colorectal tumors predict clinical outcome. Science. 2006 Sep 29;313(5795):1960-4. doi: 10.1126/science.1129139. PMID 17008531
- [Background] Galon J, Fridman WH, Pages F. The adaptive immunologic microenvironment in colorectal cancer: a novel perspective. Cancer Res. 2007 Mar 1;67(5):1883-6. doi: 10.1158/0008-5472.CAN-06-4806. PMID 17332313
- [Background] Mlecnik B, Tosolini M, Kirilovsky A, Berger A, Bindea G, Meatchi T, Bruneval P, Trajanoski Z, Fridman WH, Pages F, Galon J. Histopathologic-based prognostic factors of colorectal cancers are associated with the state of the local immune reaction. J Clin Oncol. 2011 Feb 20;29(6):610-8. doi: 10.1200/JCO.2010.30.5425. Epub 2011 Jan 18. PMID 21245428
- [Background] Pages F, Berger A, Camus M, Sanchez-Cabo F, Costes A, Molidor R, Mlecnik B, Kirilovsky A, Nilsson M, Damotte D, Meatchi T, Bruneval P, Cugnenc PH, Trajanoski Z, Fridman WH, Galon J. Effector memory T cells, early metastasis, and survival in colorectal cancer. N Engl J Med. 2005 Dec 22;353(25):2654-66. doi: 10.1056/NEJMoa051424. PMID 16371631
- [Background] Pages F, Kirilovsky A, Mlecnik B, Asslaber M, Tosolini M, Bindea G, Lagorce C, Wind P, Marliot F, Bruneval P, Zatloukal K, Trajanoski Z, Berger A, Fridman WH, Galon J. In situ cytotoxic and memory T cells predict outcome in patients with early-stage colorectal cancer. J Clin Oncol. 2009 Dec 10;27(35):5944-51. doi: 10.1200/JCO.2008.19.6147. Epub 2009 Oct 26. PMID 19858404
- [Background] Butterfield LH, Disis ML, Fox BA, Lee PP, Khleif SN, Thurin M, Trinchieri G, Wang E, Wigginton J, Chaussabel D, Coukos G, Dhodapkar M, Hakansson L, Janetzki S, Kleen TO, Kirkwood JM, Maccalli C, Maecker H, Maio M, Malyguine A, Masucci G, Palucka AK, Potter DM, Ribas A, Rivoltini L, Schendel D, Seliger B, Selvan S, Slingluff CL Jr, Stroncek DF, Streicher H, Wu X, Zeskind B, Zhao Y, Zocca MB, Zwierzina H, Marincola FM. A systematic approach to biomarker discovery; preamble to "the iSBTc-FDA taskforce on immunotherapy biomarkers". J Transl Med. 2008 Dec 23;6:81. doi: 10.1186/1479-5876-6-81. PMID 19105846
- [Background] Butterfield LH, Palucka AK, Britten CM, Dhodapkar MV, Hakansson L, Janetzki S, Kawakami Y, Kleen TO, Lee PP, Maccalli C, Maecker HT, Maino VC, Maio M, Malyguine A, Masucci G, Pawelec G, Potter DM, Rivoltini L, Salazar LG, Schendel DJ, Slingluff CL Jr, Song W, Stroncek DF, Tahara H, Thurin M, Trinchieri G, van Der Burg SH, Whiteside TL, Wigginton JM, Marincola F, Khleif S, Fox BA, Disis ML. Recommendations from the iSBTc-SITC/FDA/NCI Workshop on Immunotherapy Biomarkers. Clin Cancer Res. 2011 May 15;17(10):3064-76. doi: 10.1158/1078-0432.CCR-10-2234. Epub 2011 May 10. PMID 21558394
- [Background] Tahara H, Sato M, Thurin M, Wang E, Butterfield LH, Disis ML, Fox BA, Lee PP, Khleif SN, Wigginton JM, Ambs S, Akutsu Y, Chaussabel D, Doki Y, Eremin O, Fridman WH, Hirohashi Y, Imai K, Jacobson J, Jinushi M, Kanamoto A, Kashani-Sabet M, Kato K, Kawakami Y, Kirkwood JM, Kleen TO, Lehmann PV, Liotta L, Lotze MT, Maio M, Malyguine A, Masucci G, Matsubara H, Mayrand-Chung S, Nakamura K, Nishikawa H, Palucka AK, Petricoin EF, Pos Z, Ribas A, Rivoltini L, Sato N, Shiku H, Slingluff CL, Streicher H, Stroncek DF, Takeuchi H, Toyota M, Wada H, Wu X, Wulfkuhle J, Yaguchi T, Zeskind B, Zhao Y, Zocca MB, Marincola FM. Emerging concepts in biomarker discovery; the US-Japan Workshop on Immunological Molecular Markers in Oncology. J Transl Med. 2009 Jun 17;7:45. doi: 10.1186/1479-5876-7-45. PMID 19534815
- [Background] Bindea G, Mlecnik B, Fridman WH, Pages F, Galon J. Natural immunity to cancer in humans. Curr Opin Immunol. 2010 Apr;22(2):215-22. doi: 10.1016/j.coi.2010.02.006. Epub 2010 Mar 6. PMID 20207124
- [Background] Pages F, Galon J, Dieu-Nosjean MC, Tartour E, Sautes-Fridman C, Fridman WH. Immune infiltration in human tumors: a prognostic factor that should not be ignored. Oncogene. 2010 Feb 25;29(8):1093-102. doi: 10.1038/onc.2009.416. Epub 2009 Nov 30. PMID 19946335
- [Background] Broussard EK, Disis ML. TNM staging in colorectal cancer: T is for T cell and M is for memory. J Clin Oncol. 2011 Feb 20;29(6):601-3. doi: 10.1200/JCO.2010.32.9078. Epub 2011 Jan 18. No abstract available. PMID 21245434
- [Background] Halama N, Michel S, Kloor M, Zoernig I, Benner A, Spille A, Pommerencke T, von Knebel DM, Folprecht G, Luber B, Feyen N, Martens UM, Beckhove P, Gnjatic S, Schirmacher P, Herpel E, Weitz J, Grabe N, Jaeger D. Localization and density of immune cells in the invasive margin of human colorectal cancer liver metastases are prognostic for response to chemotherapy. Cancer Res. 2011 Sep 1;71(17):5670-7. doi: 10.1158/0008-5472.CAN-11-0268. Epub 2011 Aug 16. PMID 21846824
- [Background] Camus M, Tosolini M, Mlecnik B, Pages F, Kirilovsky A, Berger A, Costes A, Bindea G, Charoentong P, Bruneval P, Trajanoski Z, Fridman WH, Galon J. Coordination of intratumoral immune reaction and human colorectal cancer recurrence. Cancer Res. 2009 Mar 15;69(6):2685-93. doi: 10.1158/0008-5472.CAN-08-2654. Epub 2009 Mar 3. PMID 19258510
- [Background] Tesniere A, Apetoh L, Ghiringhelli F, Joza N, Panaretakis T, Kepp O, Schlemmer F, Zitvogel L, Kroemer G. Immunogenic cancer cell death: a key-lock paradigm. Curr Opin Immunol. 2008 Oct;20(5):504-11. doi: 10.1016/j.coi.2008.05.007. Epub 2008 Jun 23. PMID 18573340
- [Background] Ghiringhelli F, Menard C, Puig PE, Ladoire S, Roux S, Martin F, Solary E, Le Cesne A, Zitvogel L, Chauffert B. Metronomic cyclophosphamide regimen selectively depletes CD4+CD25+ regulatory T cells and restores T and NK effector functions in end stage cancer patients. Cancer Immunol Immunother. 2007 May;56(5):641-8. doi: 10.1007/s00262-006-0225-8. Epub 2006 Sep 8. PMID 16960692
- [Background] Machiels JP, Reilly RT, Emens LA, Ercolini AM, Lei RY, Weintraub D, Okoye FI, Jaffee EM. Cyclophosphamide, doxorubicin, and paclitaxel enhance the antitumor immune response of granulocyte/macrophage-colony stimulating factor-secreting whole-cell vaccines in HER-2/neu tolerized mice. Cancer Res. 2001 May 1;61(9):3689-97. PMID 11325840
- [Background] Mlecnik B, Tosolini M, Charoentong P, Kirilovsky A, Bindea G, Berger A, Camus M, Gillard M, Bruneval P, Fridman WH, Pages F, Trajanoski Z, Galon J. Biomolecular network reconstruction identifies T-cell homing factors associated with survival in colorectal cancer. Gastroenterology. 2010 Apr;138(4):1429-40. doi: 10.1053/j.gastro.2009.10.057. Epub 2009 Nov 10. PMID 19909745
- [Background] Branford S. Chronic myeloid leukemia: molecular monitoring in clinical practice. Hematology Am Soc Hematol Educ Program. 2007:376-83. doi: 10.1182/asheducation-2007.1.376. PMID 18024654
- [Background] Campbell PJ, Stephens PJ, Pleasance ED, O'Meara S, Li H, Santarius T, Stebbings LA, Leroy C, Edkins S, Hardy C, Teague JW, Menzies A, Goodhead I, Turner DJ, Clee CM, Quail MA, Cox A, Brown C, Durbin R, Hurles ME, Edwards PA, Bignell GR, Stratton MR, Futreal PA. Identification of somatically acquired rearrangements in cancer using genome-wide massively parallel paired-end sequencing. Nat Genet. 2008 Jun;40(6):722-9. doi: 10.1038/ng.128. Epub 2008 Apr 27. PMID 18438408
- [Background] Diehl F, Schmidt K, Choti MA, Romans K, Goodman S, Li M, Thornton K, Agrawal N, Sokoll L, Szabo SA, Kinzler KW, Vogelstein B, Diaz LA Jr. Circulating mutant DNA to assess tumor dynamics. Nat Med. 2008 Sep;14(9):985-90. doi: 10.1038/nm.1789. Epub 2007 Jul 31. PMID 18670422
- [Background] Yung TK, Chan KC, Mok TS, Tong J, To KF, Lo YM. Single-molecule detection of epidermal growth factor receptor mutations in plasma by microfluidics digital PCR in non-small cell lung cancer patients. Clin Cancer Res. 2009 Mar 15;15(6):2076-84. doi: 10.1158/1078-0432.CCR-08-2622. Epub 2009 Mar 10. PMID 19276259
- [Background] Leary RJ, Kinde I, Diehl F, Schmidt K, Clouser C, Duncan C, Antipova A, Lee C, McKernan K, De La Vega FM, Kinzler KW, Vogelstein B, Diaz LA Jr, Velculescu VE. Development of personalized tumor biomarkers using massively parallel sequencing. Sci Transl Med. 2010 Feb 24;2(20):20ra14. doi: 10.1126/scitranslmed.3000702. PMID 20371490
- [Background] McBride DJ, Orpana AK, Sotiriou C, Joensuu H, Stephens PJ, Mudie LJ, Hamalainen E, Stebbings LA, Andersson LC, Flanagan AM, Durbecq V, Ignatiadis M, Kallioniemi O, Heckman CA, Alitalo K, Edgren H, Futreal PA, Stratton MR, Campbell PJ. Use of cancer-specific genomic rearrangements to quantify disease burden in plasma from patients with solid tumors. Genes Chromosomes Cancer. 2010 Nov;49(11):1062-9. doi: 10.1002/gcc.20815. PMID 20725990